CLINICAL TRIAL: NCT05991817
Title: Study of the Effect of Sevoflurane General Anesthetic on Spatial Memory in Humans
Brief Title: Sevoflurane General Anesthetic and Spatial Memory in Humans
Status: Recruiting | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Other Study IDs: OAIC: 1328/23
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Spatial Memory Disorder
MeSH Terms: conditions — Memory Disorders | interventions — Surgical Procedures, Operative; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults 30-50 years
  Interventions: Procedure: Surgery/general anesthesia

INTERVENTIONS:
Procedure: Surgery/general anesthesia — Adult patients between the ages of 30 and 50 who are to undergo elective surgery under general anesthesia will have their spatial memory tested and interleukin 1beta and alpha tumor necrosis measured before and after surgery.

SUMMARY:
The goal of this observational study is to learn about the effect of general anesthetic on spatial memory in adults who will undergo to an elective surgery. The main question it aims to answer is:

• A surgical event under general anesthesia with sevoflurane transiently impairs spatial memory in humans and induces an increase in inflammatory cytokines.

Participants will perform a virtual maze test and plasma samples will be taken before and after surgery.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) occurs after a surgical event under general anesthesia and is characterized by a decline in one or more cognitive functions. POCD is defined as delayed neurocognitive recovery if it takes place within the first 30 days, if it exceeds that time it is known as postoperative neurocognitive disorder. The pathogenesis of this dysfunction is not entirely clear. However, the most accepted hypothesis would be neuroinflammatory, which would take place due to the contribution of inflammatory factors typical of surgical trauma under general anesthesia, with anesthetics such as sevoflurane. Consequently, one of the areas most susceptible to this inflammatory environment would be the hippocampus, a structure responsible for learning and memory. Spatial memory is responsible for encoding and retrieving information about the environment and spatial orientation. To confirm this hypothesis, an elective laparoscopic cholecystectomy under general anesthesia with sevoflurane, plasma measurement of cytokines interleukin-1beta and tumor necrosis factor-alpha and virtual navigation tests will be performed before and after an elective laparoscopic cholecystectomy under general anesthesia with sevoflurane, in order to establish a correlation between the inflammatory component and performance in the virtual navigation test. The above will allow us to elucidate the possible occurrence of a delayed neurocognitive recovery related to spatial memory in middle-aged individuals, providing new background related to an age group that has been little studied, with a non-minor incidence (30%), where the evident concern arises for being a population exposed to activities or environments of greater risk, linked to work, sport, driving, among others. This finding will guide the doctor and the patient to decide or take the necessary safeguards when proceeding with a surgical intervention in the middle-aged population.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for elective laparoscopic surgery of cholecystectomy.
* Age 30 to 50 years.

Exclusion Criteria:

* Visual or hearing difficulties.
* Malignant hyperthermia.
* Being treated with centrally acting drugs, such as anxiolytics, antidepressants, antipsychotics, anticonvulsants, anticholinergics, and first-generation antihistamines.
* Present a disorder of the sphere of neuropsychiatry
* Substance abuse disorder.

Ages: 30 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Adult patients bewteen 30 and 50 years old who will undergo to an elective laparoscopic surgery of cholecystectomy.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Virtual spatial memory | 1th day after surgery
  Time to reach the goal

SECONDARY OUTCOMES:
Interleukin-1beta | 1st day after surgery
  Interleukin-1beta plasma concentration
Interleukin-1beta | 7th day after surgery
  Interleukin-1beta plasma concentration
Interleukin-1beta | 30th day after surgery
  Interleukin-1beta plasma concentration
Tumor necrosis factor alpha | 1st day after surgery
  Tumor necrosis factor alpha plasma concentration
Tumor necrosis factor alpha | 7th day after surgery
  Tumor necrosis factor alpha plasma concentration
Tumor necrosis factor alpha | 30th day after surgery
  Tumor necrosis factor alpha plasma concentration
Virtual spatial memory | 7st day after surgery
  Time to reach the goal
Virtual spatial memory | 30th day after surgery
  Time to reach the goal

CONTACTS AND LOCATIONS:
Overall Officials: Khaleed Etchegaray, Principal Investigator — University of Chile; Jamileth More, PhD, Study Director — University of Chile; Antonello Penna, MD, PhD, Study Director — University of Chile
Locations (2):
- Chile (2):
  - Centro de Investigación Cínica Avanzada (CICA), Hospital Clinico de la Universidad de Chile, Santiago, RM
  - Hospital Clinico de la Universidad de Chile, Santiago, RM

IPD SHARING:
Plan to Share IPD: Undecided